CLINICAL TRIAL: NCT05063643
Title: Cardiotoxicity of Targeted Therapy for HER-2 Positive Breast Cancer Patients at High altitude-a Multicenter, Prospective Cohort Study
Brief Title: Cardiotoxicity of Targeted Therapy for HER-2 Positive Breast Cancer Patients at High Altitude
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Affiliated Hospital of Qinghai University (Other)
Responsible Party: Principal Investigator, Jiuda Zhao, Professor, Affiliated Hospital of Qinghai University
Other Study IDs: SL-2020076
Record Dates: First submitted 2021-07-26; First posted 2021-10-01 (Actual); Last update posted 2021-10-01 (Actual); Status verified 2021-09

CONDITIONS: HER2-positive Breast Cancer; Targeted Therapy; Cardiac Toxicity; High Altitude
Keywords: HER2-positive breast cancer; Targeted therapy; Cardiotoxicity; High Altitude
MeSH Terms: conditions — Cardiotoxicity; Altitude Sickness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: High altitude — High altitude is defined as >2000m.

SUMMARY:
This is a prospective, multicenter, cohort study aiming to explore the cardiotoxicity of targeted therapy for HER-2 positive breast cancer patients who lives in high altitude area. One hundred and thirty two HER-2 positive breast cancer patients who will receive neoadjuvant, adjuvant, or palliative targeted therapy will be enrolled. The cardiotoxicity of targeted therapy will be observed and recorded during the treatment and one year after the end of treatment. The subjects will be stratified by age, baseline cardiac risk factors, and anthracyclines.

DETAILED DESCRIPTION:
HER-2 positive breast cancer patients who live at high altitudes greater than 2000 meters for long periods of time and will receive trastuzumab-based targeted therapy will be enrolled. The subjects included early and advanced patients. Treatment regimens includes chemotherapy combined with trastuzumab, chemotherapy combined with trastuzumab and pertuzumab, trastuzumab alone, and trastuzumab plus pertuzumab. Electrocardiogram, cardiac ultrasound, NT-proBNP, and TNI will be tested every 3 months when the treatment begins. The primary endpoint is cardiotoxity. The second endpoints is pathologic complete response (pCR) rate in neoadjuvant therapy, objective remission rate (ORR) and disease control rate (DCR) in neoadjuvant and palliative therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed invasive HER2-positive breast cancer.
2. The baseline left ventricular ejection fraction >55%.
3. Living at high altitude area （>2000 meters）for at least 10 years.
4. ECOG score 0-2.
5. Expected survival time ≥ 12 months.

Exclusion Criteria:

1. Patients with previous breast cancer or other malignant tumor within 5 years.
2. Patients who had accepted previous anti-HER2 or anthracyclines-based therapy.
3. Patients with severe heart disease or discomfort.
4. Patients who are pregnant.
5. Patients with other conditions considered not suitable to be enrolled by the investigator.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All enrolled patients are from four centers of Qinghai province.
Sampling Method: Non-Probability Sample
Enrollment: 132 (Estimated)
Dates: Start 2021-10 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Incidence rate of cardiotoxicity | 5 years
  Cardiotoxicity includes death from cardiac cause, severe congestive heart failure (New York Heart Association Class III or IV), more than 10% decrease of left ventricular ejection fraction (LVEF) and to below 50%, and an asymptomatic or mildly symptomatic (NYHA class II) substantial decrease in LVEF.

SECONDARY OUTCOMES:
pCR rate | 4 years
  Pathologic complete response (pCR) rate in patients received neoadjuvant therapy
ORR | 4 years
  Objective remission rate in patients received neoadjuvant and palliative therapy
DCR | 4 years
  Disease control rate in patients received neoadjuvant and palliative therapy
OS | 5 years
  Overall survival of the enrolled patients
the incidence of treatment-related adverse events | 5 years
  Incidence and Severity of adverse events according to the CTC AE V4.03 Incidence and Severity of adverse events according to the CTC AE V4.03 Incidence and severity of adverse events according to the CTC AE V4.03

CONTACTS AND LOCATIONS:
Locations (1):
- Affiliated Hospital of Qinghai University, Xining, Qinghai, China